CLINICAL TRIAL: NCT05666297
Title: Screening of Cardiac Abnormalities in the First Trimester of Pregnancy by Volumetric Acquisition: an International Multicenter Study
Brief Title: Screening of Cardiac Abnormalities in the First Trimester of Pregnancy by Volumetric Acquisition
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Antonio Schiattarella, MD, University of Campania Luigi Vanvitelli
Other Study IDs: 37885
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy; Ultrasound; Fetal Conditions; Cardiac Abnormalities
Keywords: pregnancy; ultrasound; fetal abnormalities; Cardiac Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ultrasound is one of the most important tools in pregnancy both for its diagnostic capacity, but also because it is not invasive.

For physiological pregnancy, the Italian guidelines provide for the execution of 3 ultrasounds: one in the first trimester (between 11 and 14 weeks), one in the second trimester (between 20 and 22 weeks) and one in the third (between 30 and 36 weeks). weeks).

Screening for cardiac abnormalities is done during second trimester ultrasound, also called structural ultrasound. However, the development of three-dimensional (3D) sonography has represented a dramatic shift in obstetrics as it allows for the acquisition of a volume of data rather than conventional planar or 2D scans. This method has allowed considerable progress in the study of the fetus in the initial stages of development and has opened new windows in the knowledge of anatomical malformations at an early age.

The possibility of detecting structural anomalies already during the first trimester of pregnancy allows, in fact, to provide the patient with additional time for counseling and for any genetic tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the obstetric ultrasound clinic for the execution of the first trimester ultrasound between 11+0 and 13+6 weeks of gestation

Exclusion Criteria:

* Less than 18 years old
* Multiple gestations
* Women with an altered state of consciousness, seriously ill, with mental handicaps;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study in question will be conducted prospectively at the structures involved. Participation in the study will be offered to all patients referred to the obstetric ultrasound clinic for the execution of the first trimester ultrasound between 11+0 and 13+6 weeks of gestation, foreseen in normal clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiac abnormalities found in the first trimester of pregnancy | Between 11+0 and 13+6 days of pregnancy
  Incidence of cardiac abnormalities found in the first trimester of pregnancy by 3D scan

SECONDARY OUTCOMES:
Gestational age at delivery | delivery
  Weeks of gestation at the moment of delivery
Preterm birth rates | Less than 24, 28, 34 weeks gestation
Birth weight | delivery
  Weight of the baby at the time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Fabiana Savoia, MD, Study Chair — University of Campania Luigi Vanvitelli; Antonio Schiattarella, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy